CLINICAL TRIAL: NCT06805747
Title: A Comparative Study of Ventilation Strategies in Different Surgical Positions on Intracranial Pressure and Cerebral Blood Flow During Laparoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inner Mongolia Baogang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-MER-312
Record Dates: First submitted 2025-01-19; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Laparoscopic Surgery
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- T-V-VCV Group (Experimental): Variable tidal volume ventilation (V-VCV) ：The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 41%.
  Use of the trendelenburg position：Lower the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Variable tidal volume ventilation (V-VCV); Other: Trendelenburg position
- T-PRVC Group (Experimental): Pressure-regulated volume-controlled ventilation (PRVC) ：The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW), the upper limit of peak inspiratory pressure was 30 cmH2O, the maximum tidal volume (Vt_max) and the minimum tidal volume (Vt_min) was set at 10-20% of the base tidal volume (Vt_base). Respiratory Rate is 12, Inspiration to Expiration Ratio is 1:2, Positive End-Expiratory Pressure (PEEP) is 5cmH2O, and Inhaled Oxygen Concentration (FiO2) is 98%.
  Use of the trendelenburg position：Lower the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Pressure-regulated volume-controlled ventilation (PRVC); Other: Trendelenburg position
- T-C-VCV Group (Experimental): Conventional volume-controlled ventilation (C-VCV)The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12.Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 98%.
  Use of the trendelenburg position：Lower the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Conventional volume-controlled ventilation (C-VCV); Other: Trendelenburg position
- T-PVC Group (Experimental): Pressure-controlled ventilation (PCV)：The inspiratory pressure level is set, usually with an initial value of 20 cmH2O, a respiratory rate of 12, an inspiratory/expiratory ratio of 1:2, a positive end-expiratory pressure (PEEP) of 5 cm water column, and an inspired oxygen concentration (FiO2) of 98%.
  Use of the trendelenburg position：Lower the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Pressure-controlled ventilation (PCV); Other: Trendelenburg position
- R-V-VCV Group (Experimental): Variable tidal volume ventilation (V-VCV) ：The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 41%.
  Use of the reverse trendelenburg position：Elevate the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Variable tidal volume ventilation (V-VCV); Other: Reverse Trendelenburg position
- R-PRVC Group (Experimental): Pressure-regulated volume-controlled ventilation (PRVC) ：The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW), the upper limit of peak inspiratory pressure was 30 cmH2O, the maximum tidal volume (Vt_max) and the minimum tidal volume (Vt_min) was set at 10-20% of the base tidal volume (Vt_base). Respiratory Rate is 12, Inspiration to Expiration Ratio is 1:2, Positive End-Expiratory Pressure (PEEP) is 5cmH2O, and Inhaled Oxygen Concentration (FiO2) is 98%.
  Use of the reverse trendelenburg position：Elevate the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Pressure-regulated volume-controlled ventilation (PRVC); Other: Reverse Trendelenburg position
- R-C-VCV Group (Experimental): Conventional volume-controlled ventilation (C-VCV)The initial tidal volume was set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW).The maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) were set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12.Inspiratory Flow Rate (IFR) 60L/min, Inspiratory to Expiratory Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, and Inhaled Oxygen Concentration (FiO2) 98%.
  Use of the reverse trendelenburg position：Elevate the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Conventional volume-controlled ventilation (C-VCV); Other: Reverse Trendelenburg position
- R-PVC Group (Experimental): Pressure-controlled ventilation (PCV)：The inspiratory pressure level is set, usually with an initial value of 20 cmH2O, a respiratory rate of 12, an inspiratory/expiratory ratio of 1:2, a positive end-expiratory pressure (PEEP) of 5 cm water column, and an inspired oxygen concentration (FiO2) of 98%.
  Use of the reverse trendelenburg position：Elevate the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Interventions: Other: Pressure-controlled ventilation (PCV); Other: Reverse Trendelenburg position

INTERVENTIONS:
Other: Variable tidal volume ventilation (V-VCV) — Variable tidal volume ventilation (V-VCV) ：The initial tidal volume is set at 6-8 ml/kg IBW according to the Ideal Body Weight (IBW), and the maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) are set at 10-20% of the base tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiration to Expiration Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5 cm water column, and Inhaled Oxygen Concentration (FiO2) 41%.
  Arms: R-V-VCV Group; T-V-VCV Group
Other: Pressure-regulated volume-controlled ventilation (PRVC) — Pressure-regulated volume-controlled ventilation (PRVC) ：Initial tidal volume is set at 6-8 ml/kg IBW based on Ideal Body Weight (IBW), peak inspiratory pressure is capped at 30 cmH2O, maximum tidal volume (Vt_max), and minimum tidal volume (Vt_min) is set at 10-20% of basal tidal volume (Vt_base). Respiratory Rate (RR) 12, Inspiratory Breathing Ratio (IBR) 1:2, Positive End-Expiratory Pressure (PEEP) 5 cm water column, and Inhaled Oxygen Concentration (FiO2) 98%.
  Arms: R-PRVC Group; T-PRVC Group
Other: Conventional volume-controlled ventilation (C-VCV) — Conventional volume-controlled ventilation (C-VCV) ：The initial tidal volume is set at 6-8 ml/kg IBW based on Ideal Body Weight (IBW), and the maximum tidal volume (Vt_max) and minimum tidal volume (Vt_min) are set at 10-20% of the basal tidal volume (Vt_base). Respiratory Rate 12. Inspiratory Flow Rate (IFR) 60L/min, Inspiration to Expiration Ratio (IER) 1:2, Positive End-Expiratory Pressure (PEEP) 5cm water column, FiO2 98%.
  Arms: R-C-VCV Group; T-C-VCV Group
Other: Pressure-controlled ventilation (PCV) — Pressure-controlled ventilation (PCV)：Set inspiratory pressure level, usually 20 cmH2O initial value, Respiratory Rate 12, Inspiratory to Expiratory Ratio 1:2, Positive End-Expiratory Pressure (PEEP) 5 cm water column, Inhaled Oxygen Concentration (FiO2) 98%.
  Arms: R-PVC Group; T-PVC Group
Other: Trendelenburg position — Trendelenburg position：Lower the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Arms: T-C-VCV Group; T-PRVC Group; T-PVC Group; T-V-VCV Group
Other: Reverse Trendelenburg position — Reverse Trendelenburg position：Elevate the head of the bed by 30 degrees with no more than 15 degrees of lateral tilt.
  Arms: R-C-VCV Group; R-PRVC Group; R-PVC Group; R-V-VCV Group

SUMMARY:
The purpose of this clinical trial is to investigate the effects of laparoscopic surgery in the Trendelenburg and Reverse Trendelenburg positions, and variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), and pressure-controlled ventilation (PCV) on esophageal pressure, airway pressure, tidal volume, intracranial pressure, and cerebral blood flow.

The study aims to address the following primary questions:Does laparoscopic surgery in the Trendelenburg or Reverse Trendelenburg position increase esophageal pressure, airway pressure, and intracranial pressure, and decrease tidal volume and cerebral blood flow? Do variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), or pressure-controlled ventilation (PCV) increase esophageal pressure, airway pressure, and intracranial pressure, and decrease tidal volume and cerebral blood flow? The investigators will compare variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), and pressure-controlled ventilation (PCV) to determine which ventilation mode results in the least physiological disturbance for patients.

Participant Procedures:

Participants will: Be positioned according to the surgical requirements.Be randomly assigned to mechanical ventilation with either variable tidal volume ventilation (V-VCV), pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), or pressure-controlled ventilation (PCV).

Undergo assessments at the following time points: immediately after endotracheal intubation, immediately after pneumoperitoneum, immediately after position change (Trendelenburg or Reverse Trendelenburg), 30 minutes after position change, and 1 hour after position change.

Have their esophageal pressure, airway pressure, intracranial pressure, tidal volume, and internal jugular vein blood flow recorded at each assessment time point.

ELIGIBILITY:
Inclusion Criteria:

* Age: Unrestricted
* American Society of Anesthesiologists (ASA) Physical Status: Class I-III
* Surgical Position: Requires the use of either the Trendelenburg position or the Reverse Trendelenburg position during the procedure.
* Ventilation: Planned mechanical ventilation is required during the procedure, with suitability for one of the following modes: pressure-regulated volume-controlled ventilation (PRVC), conventional volume-controlled ventilation (C-VCV), or pressure-controlled ventilation (PCV).

Exclusion Criteria:

* Significant Cardiopulmonary Disease:
* Intracranial Disease
* Severe Coagulopathy or Current Anticoagulant Therapy
* Presence of Psychiatric Illness, Cognitive Impairment, or other condition that precludes the ability to understand or comply with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
esophageal pressure | immediately after tracheal intubation
airway pressure | immediately after tracheal intubation
intracranial pressure | immediately after pneumoperitoneum
tidal volume | immediately after tracheal intubation
carotid blood flow | half an hour after change of position

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: January 2026-January 2036
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.